CLINICAL TRIAL: NCT02535455
Title: Development and Pilot of Positive Self-Reappraisal Emotion Regulation Intervention to Improve Self-Care Among HIV+ Substance Users
Brief Title: Acceptance and Compassion to Enhance Self-care Pilot
Acronym: ACES Pilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: A118121
Record Dates: First submitted 2015-08-20; First posted 2015-08-28 (Estimated); Last update posted 2020-06-19 (Actual); Status verified 2020-06

CONDITIONS: HIV/AIDS; Substance Use Disorder
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ACES Pilot (Experimental): This pilot will consist of 5 individual sessions and an innovative bi-directional text message component that uses participant-written positive self-statements informed by the intervention content (e.g., self-compassion, positive self-reappraisal and nonjudgmental acceptance).
  Interventions: Behavioral: ACES Pilot

INTERVENTIONS:
Behavioral: ACES Pilot — This pilot will consist of 5 individual sessions and an innovative bi-directional text message component that uses participant-written positive self-statements informed by the intervention content (e.g., self-compassion, positive self-reappraisal and nonjudgmental acceptance).
  Other Names: Acceptance and Compassion to Enhance Self-care

SUMMARY:
Innovative approaches are needed to optimize the benefits of treatment as prevention (TasP) among HIV+ substance users, who experience profound health disparities that amplify onward transmission risk. This project will systematically develop, refine and conduct an open pilot to assess the feasibility and acceptability of a two-phase emotion regulation intervention that targets emotional barriers to HIV-related self-care among individuals who endorse active substance use. Emotional barriers such as shame and internalized stigma have been identified as barriers to optimal HIV care among individuals struggling with HIV and substance use. To effectively implement TasP, strategies for addressing these barriers are needed. Utilizing transdiagnostic approaches (e.g., positive affect-focused emotional regulation, mindfulness and self-compassion) investigators will develop, refine and pilot a two-phase emotional regulation intervention that requires only 5 face-to-face hours and can ultimately be implemented by a case-management-level staff person or trained peer educator. The first phase of the intervention will be a multicomponent in-person intervention targeting emotional, cognitive and behavioral barriers to HIV self-care behaviors among HIV+ substance users. The second phase of the intervention will extend the intervention benefits by sending personalized positive self-reappraisal text messages in response to text message queries about participants' mood. This phase will use an innovative personalized bi-directional platform, which will leverage an existing text message delivery system. This project will be instrumental in developing a relatively low-resource intervention strategy to address unmet emotional barriers to optimal HIV-care among individuals who are actively using substances. This work will provide the necessary pilot data for a subsequent grant submission to assess the preliminary efficacy of the intervention. The resulting intervention has the potential to address emotional barriers to self-care along the HIV care cascade: including retention in care, antiretroviral treatment adherence and persistence, and ultimately viral suppression.

DETAILED DESCRIPTION:
Investigators will develop and refine a two-phase emotion regulation intervention. This process will involve 5 steps: 1) conducting 5-8 key informant interviews, including obtaining feedback on a drafted manual and materials from providers and case managers, 2) integrating the qualitative data, 3) running 2 participants through a condensed version of the intervention and obtaining feedback on the content, language, and text message interface, 4) integrating the additional feedback, and 5) conducting an open pilot with 10 participants to assess feasibility and acceptability of the revised intervention. The pilot will include 3 research assessment visits which will involve completion of self-report questionnaires using Qualtrics at baseline, within one week of completion of phase 1, and within one week of completing phase 2. Viral load (VL) will be assessed at baseline and at the final follow up.

Qualitative interviews. The investigators will conduct 5-8 semi-structured qualitative interviews with providers and case managers. Interviews will inquire about unmet psychological barriers to HIV-care, perceptions of proposed domains and text message questions and response options. All interviews will be recorded, transcribed and analyzed using thematic analysis. Prominent themes and suggestions brought up in the interviews will be integrated into the intervention materials and implementation.

Trial run of pilot. After integrating the feedback from the key informant interviews, investigators will recruit two participants to complete a condensed version of the intervention. After each of the 5 sessions, participants will be asked to complete perceived usefulness surveys. Both participants will then be interviewed to obtain feedback on the intervention. These interviews will be recorded, transcribed and analyzed using thematic analysis. Prominent themes and suggestions brought up in these interviews as well as logistic challenges will be integrated into the intervention materials and implementation procedures.

Text messages. Investigators will use questions adapted from a previously published personalized bi-directional text message intervention involving HIV+ substance users (TxText) to assess mood, adherence and substance use. Each participant will receive 3 texts/week inquiring about current mood over the course of the intervention. Additionally, in phase 2 each participant will receive weekly texts asking about their medication adherence. Given the stigmatized nature of substance use, investigators will use a coded query, adapted from TxText, which assess substance use in the form of a weather question. This coded query strategy has demonstrated feasibility and acceptability among a similar population of HIV+ active substance users. All participants will be reminded of the meaning of this question during phase 1. During the last in-person intervention visit, participants will identify 5 positive self-reappraisal statements and link them to response options to the mood query based on when they feel each would be most helpful in regulating their emotions. Throughout phase 2, participants will then receive their linked positive-self reappraisal statements in response to mood queries. Participants will then be asked to respond on a 6-point scale indicating how helpful the positive self-reappraisal was (0=extremely unhelpful to 5= extremely helpful), which will be used to assess engagement in phase 2 of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking
* HIV+
* ≥18 years old
* Able to complete informed consent
* Endorse polysubstance use in the past 2 months, excluding cannabis and tobacco
* Participants must own a cell phone with text message capacity and be willing to work with a study staff member to add minutes or money to their cell phone plan to cover the text-message component of the intervention (at no cost to participants).
* Consent to release their medical records, in order to assess engagement in HIV-care (i.e., attended/scheduled appointments).

Exclusion Criteria:

* Endorsement of active suicidality or psychosis on initial clinical interview.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-08-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline antiretroviral adherence to post intervention follow up visits | Collected at baseline, research visit after face-to-face intervention component (approximately 5 weeks post-baseline) and research visit after text-message component (approximately 13 months post-baseline).
  Participants will be asked to complete the Visual Analogue Scale (VAS) in person at baseline and subsequent research visits.
Change from baseline engagement in HIV-related Care (number of HIV-related health visits scheduled and attended) to follow up visits. | Collected at baseline, research visit after face-to-face intervention component (approximately 5 weeks post-baseline) and research visit after text-message component (approximately 13 months post-baseline).
  Participants will be asked to report the number of HIV-related health visits scheduled and attended. Additionally, chart reviews will be conducted at the end of the study to determine the number of attended compared to scheduled HIV-related health visits.

SECONDARY OUTCOMES:
Change from baseline viral load to final follow up visit. | Collected at baseline and approximately 21 months post-baseline at final research visit.
  Participants will have blood drawn for viral load tests at baseline and their final follow up visit. The values will be compared.
Change in substance use | Assessed at baseline, approximately 5 weeks post-baseline, approximately 13 months post-baseline and approximately 21 months post-baseline.
  The ASSIST measures substance use.
Change in baseline sexual risk behaviors to research visit after face-to-face intervention component (approximately 5 weeks post-baseline) and research visit after text-message component (approximately 11 months post-baseline). | ssessed at baseline, approximately 5 weeks post-baseline, approximately 13 months post-baseline and approximately 21 months post-baseline.
  Self-report questions to assess recent sexual risk behaviors.
Change in HIV and Abuse Related Shame (HARSI) | Assessed at baseline, approximately 5 weeks post-baseline, approximately 13 months post-baseline and approximately 21 months post-baseline.
  The HARSI is a self report measure that assesses HIV and abuse related shame
Change in depression (CES-D) | Assessed at baseline, approximately 5 weeks post-baseline, approximately 13 months post-baseline and approximately 21 months post-baseline.
  The CES-D will be used to assess self-reported depressive symptoms
Change in Self-Compassion (Self-Compassion Scale) | Assessed at baseline, approximately 5 weeks post-baseline, approximately 13 months post-baseline and approximately 21 months post-baseline.
  The Self-Compassion Scale will be used to assess self-reported self compassion
Change in mindfulness (Five Facet Mindfulness Questionnaire) | Assessed at baseline, approximately 5 weeks post-baseline, approximately 13 months post-baseline and approximately 21 months post-baseline.
  The Five Facet Mindfulness Questionnaire will be use to assess self-reported mindfulness

CONTACTS AND LOCATIONS:
Overall Officials: Abigail W Batchelder, PhD, MPH, Principal Investigator — University of California, San Francisco